CLINICAL TRIAL: NCT00785772
Title: A Post-Marketing Clinical Pharmacokinetics Study Of Gabapentin In Japanese Epileptic Subjects With Renal Impairment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9451169
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2011-10

CONDITIONS: Renal Impairment
Keywords: Gabapentin Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: Patients with Cleatinine Clearance (CLcr) 5-14 mL/min (Experimental)
  Interventions: Drug: Gabapentin
- 2: Patients with CLcr 15-29 mL/min (Experimental)
  Interventions: Drug: Gabapentin
- 3: Patients with CLcr 30-59 mL/min (Experimental)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — 100-200mg once a day
  Arms: 1: Patients with Cleatinine Clearance (CLcr) 5-14 mL/min
Drug: Gabapentin — 200-500mg once a day
  Arms: 2: Patients with CLcr 15-29 mL/min
Drug: Gabapentin — 400-1000mg (200-500 mg twice a day)
  Arms: 3: Patients with CLcr 30-59 mL/min

SUMMARY:
The primary objectives of this study are to evaluate the pharmacokinetics (PK) following administration of gabapentin in Japanese epileptic patients with renal impairment to confirm if there are any clinically relevant differences between the plasma gabapentin concentration simulated by population PK model, which was used for the evidence of the dose adjustment for the patients with renal impairment, and observed plasma gabapentin concentration.

DETAILED DESCRIPTION:
Only one subject was able to be enrolled. Given enrollment challenges to identify additional appropriate subjects, discussion was held with the Japan Pharmaceuticals and Medical Devices Agency (PMDA) and it was agreed with the PMDA to terminate this study. The study was terminated on December 14, 2010. The study was not terminated due to any safety findings.

ELIGIBILITY:
Inclusion Criteria:

* Japanese epilepsy patients with renal impairment

Exclusion Criteria:

* NA

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Saijyo-shi, Ehime, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451169&StudyName=A%20Post-Marketing%20Clinical%20Pharmacokinetics%20Study%20Of%20Gabapentin%20In%20Japanese%20Epileptic%20Subjects%20With%20Renal%20Impairment

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date and Completion Dates: 16 March 2010 to 1 April 2010 Study Center: 1 center in Japan
Pre-assignment Details: A subject who had already been taking gabapentin was enrolled in the study.
Groups:
- Gabapentin: The dosage regimens were adjusted depending on the creatinine clearance. Duration of observation was 15 days from screening if the subject had already been treated with gabapentin and 28 days from screening if the subject was treated with gabapentin for the first time.
  The subject enrolled was on hemodialysis, receiving a maintenance dose of 300 mg twice daily for 15 days.
Period: Overall Study
Arm/Group | Gabapentin
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gabapentin
Number analyzed (Participants) | 1
Age, Customized [Number; unit: Participant]
  <=19 years | 0
  20-64 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Observed Plasma Gabapentin Concentration
Description: Plasma gabapentin concentrations were measured on Day 8 and Day 15
Time Frame: Days 8 and 15
Population: The Pharmacokinetics (PK) concentration analysis population is defined as all subjects treated who have at least 1 of the PK parameters of interest.
Measure: Mean (Full Range); unit: µg/mL
Arm/Group | Gabapentin
Number analyzed (Participants) | 1
µg/mL
  Day 8 | 38.40 [38.40 to 38.40]
  Day 15 | 44.64 [44.64 to 44.64]

2. Primary Outcome: Ratio of Observed Plasma Gabapentin Concentration to Predicted Plasma Gabapentin Concentration Based on Population Pharmacokinetics Model
Description: Ratio of observed plasma gabapentin concentration to predicted plasma gabapentin concentration based on population pharmacokinetics model were calculated on Day 8 and Day 15, respectively.
Time Frame: Days 8 and 15
Population: as for outcome 1
Measure: Number; unit: Ratio
Arm/Group | Gabapentin
Number analyzed (Participants) | 1
Ratio
  Day 8 | 2.16
  Day 15 | 2.59

3. Primary Outcome: Ratio of Observed Plasma Gabapentin Concentration to Individual Predicted Plasma Gabapentin Concentration
Description: Ratio of observed plasma gabapentin concentration to individual predicted plasma gabapentin concentration were calculated on Day 8 and Day 15, respectively.
Time Frame: Days 8 and 15
Population: as for outcome 1
Measure: Number; unit: Ratio
Arm/Group | Gabapentin
Number analyzed (Participants) | 1
Ratio
  Day 8 | 1.15
  Day 15 | 1.37

ADVERSE EVENTS:
Time Frame: From Day -7 (informed consent) until 28 days after the end of study treatment
Arm/Group | Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was completed with an enrollment of 1 subject because prolongation of the study period or a change in the inclusion criteria (the upper limit of age was deleted) did not lead to further enrollment of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.